CLINICAL TRIAL: NCT00974974
Title: A Study To Evaluate The Safety And Efficacy Of IPX066 In Advanced Parkinson's Disease
Brief Title: A Study To Evaluate The Safety And Efficacy Of IPX066 In Advanced Parkinson's Disease (ADVANCE-PD).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPX066-B09-02
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2017-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPX066 (Experimental): Following IR CD-LD dose adjustment and conversion to IPX066, subjects were assigned to Investigational product IPX066.
  Interventions: Drug: IPX066; Drug: IR CD-LD
- IR CD-LD (Active Comparator): Following IR CD-LD dose adjustment and conversion to IPX066, subjects were assigned to Investigational product IR CD-LD (active comparator).
  Interventions: Drug: IPX066; Drug: IR CD-LD

INTERVENTIONS:
Drug: IPX066 — extended-release carbidopa-levodopa capsules
  Other Names: ER CD-LD
Drug: IR CD-LD — immediate-release carbidopa-levodopa tablets
  Other Names: immediate-release carbidopa-levodopa

SUMMARY:
This is a study to evaluate the safety and efficacy of IPX066 in advanced Parkinson's disease.

DETAILED DESCRIPTION:
A randomized, double-blind, active-control, parallel-group 13-week comparison of IPX066 versus regular carbidopa-levodopa (CD-LD). Prior to randomization, subjects on a stable regular LD regimen will enter a 3-week dose-adjustment period for IR CD-LD, followed by a 6-week dose-conversion period to IPX066.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with idiopathic PD.
2. At least 30 years old at the time of PD diagnosis.
3. Currently being treated with IR LD (CD-LD or benserazide-LD) and on a stable regimen of IR LD for at least 4 weeks and:

   * Requiring a total daily IR LD dose of at least 400 mg
   * Having a minimum dosing frequency of four times per day.
4. Able to differentiate "on" state from "off" state.
5. Have predictable "off" periods.
6. Amantadine, anticholinergics, selective monoamine oxidase (MAO) type B inhibitors (e.g., selegiline, rasagiline) or dopamine agonists are allowed as long as the doses and regimens have been stable for at least 4 weeks prior to Screening and the therapy is intended to be constant throughout the course of the study.
7. Agrees to use a medically acceptable method of contraception throughout the study and for 1 month afterward.

Exclusion Criteria:

1. Diagnosed with atypical Parkinsonism or any known secondary Parkinsonian syndrome.
2. Nonresponsive to LD therapy.
3. Prior functional neurosurgical treatment for PD (e.g., ablation or deep brain stimulation) or if such procedures are anticipated during study participation.
4. Received within 4 weeks or planning to take during participation in the clinical study: any controlled-release LD product, additional CD (e.g., Lodosyn®) or benserazide (e.g. Serazide®), catechol-O-methyl transferase inhibitors (e.g., entacapone and tolcapone), nonselective MAO inhibitors, apomorphine, and antipsychotics including neuroleptic agents for the purpose of treating psychosis or bipolar disorder.
5. Allergic to Yellow Dye #5 (tartrazine).
6. History of or currently active psychosis.
7. Active or prior medical conditions such as peptic ulcers or prior surgical (e.g., bowel) procedures that would interfere with LD absorption.
8. Active or history of narrow-angle glaucoma.
9. A history of malignant melanoma or a suspicious undiagnosed skin lesion.
10. History of myocardial infarction with residual atrial, nodal, or ventricular arrhythmias, upper gastrointestinal hemorrhage, or neuroleptic malignant syndrome and/or nontraumatic rhabdomyolysis.
11. Received any investigational medications during the 4 weeks prior to Screening.
12. Unable to swallow large pills (e.g., large vitamin pills).
13. Pregnant or breastfeeding.
14. Subjects who are unable to complete a symptom diary.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (73):
- United States (35):
  - Investigator 17, Birmingham, Alabama
  - Investigator 49, Phoenix, Arizona
  - Investigator 7, Little Rock, Arkansas
  - Investigator 3, La Jolla, California
  - Investigator 31, Sunnyvale, California
  - Investigator 6, Torrance, California
  - Investigator 51, Aurora, Colorado
  - Investigator 10, New Haven, Connecticut
  - Investigator 64, Bradenton, Florida
  - Investigator 61, Hollywood, Florida
  - Investigator 5, Ocala, Florida
  - Investigator 15, Port Charlotte, Florida
  - Investigator 8, Port Charlotte, Florida
  - Investigator 4, St. Petersburg, Florida
  - Investigator 46, Augusta, Georgia
  - Investigator 38, Boise, Idaho
  - Investigator 19, Chicago, Illinois
  - Investigator 40, Chicago, Illinois
  - Investigator 39, Des Moines, Iowa
  - Investigator 29, Kansas City, Kansas
  - Investigator 1, Bingham Farms, Michigan
  - Investigator 21, New Brunswick, New Jersey
  - Investigator 25, Albany, New York
  - Investigator 8, Commack, New York
  - Investigator 12, New York, New York
  - Investigator 11, Durham, North Carolina
  - Investigator 9, Raleigh, North Carolina
  - Investigator 20, Cincinnati, Ohio
  - Investigator 42, Toledo, Ohio
  - Investigator 60, Tulsa, Oklahoma
  - Investigator 14, Charleston, South Carolina
  - Investigator 16, Dallas, Texas
  - Investigator 13, Houston, Texas
  - Investigator 65, Tacoma, Washington
  - Investigator 2, Milwaukee, Wisconsin
- Canada (3):
  - Investigator 24, London, Ontario
  - Investigator 18, Ottawa, Ontario
  - Investigator 26, Québec, Quebec
- France (5):
  - Investigator 32, Strasbourg, Alsace
  - Investigator 22, Dijon, Bourgogne-Franche-Comté
  - Investigator 52, Lille, Hauts-de-France
  - Investigator 33, Toulouse, Midi-pyrenees
  - Investigator 58, Paris, Île-de-France Region
- Germany (6):
  - Investigator 30, Sachsen, Dresden
  - Investigator 27, Westerstede, Lower Saxony
  - Investigator 23, Berlin
  - Investigator 72, Berlin
  - Investigator 28, Berlin
  - Investigator 67, Berlin
- Poland (7):
  - Investigator 48, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigator 37, Krakow, Lesser Poland Voivodeship
  - Investigator 59, Lublin, Lublin Voivodeship
  - Investigator 36, Warsaw, Masovian Voivodeship
  - Investigator 54, Szczecin, West Pomeranian Voivodeship
  - Investigator 35, Mosina, Wielkopoloskie
  - Investigator 34, Katowice
- Romania (4):
  - Investigator 69, Târgu Mureş, Mureș County
  - Investigator 68, Brasov
  - Investigator 62, Bucharest
  - Investigator 63, Târgu Mureş
- Spain (6):
  - Investigator 43, Terrassa, Barcelona
  - Investigator 70, Barcelona
  - Investigator 57, Barcelona
  - Investigator 45, Barcelona
  - Investigator 50, Madrid
  - Investigator 53, Madrid
- Ukraine (7):
  - Investigator 55, Dnipro, Dnipropetrovsk Oblast
  - Investigator 56, Vinnitsa, Vinnytsya
  - Investigator 47, Zaporizhzhya, Zaporizhzhya
  - Investigator 71, Donetsk
  - Investigator 44, Kharkiv
  - Investigator 66, Odesa
  - Investigator 41, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morgan JC, Dhall R, Rubens R, Khanna S, Gupta S. Dosing Patterns during Conversion to IPX066, Extended-Release Carbidopa-Levodopa (ER CD-LD), in Parkinson's Disease with Motor Fluctuations. Parkinsons Dis. 2018 Oct 22;2018:9763057. doi: 10.1155/2018/9763057. eCollection 2018. PMID 30425824
- [Derived] Hauser RA, Hsu A, Kell S, Espay AJ, Sethi K, Stacy M, Ondo W, O'Connell M, Gupta S; IPX066 ADVANCE-PD investigators. Extended-release carbidopa-levodopa (IPX066) compared with immediate-release carbidopa-levodopa in patients with Parkinson's disease and motor fluctuations: a phase 3 randomised, double-blind trial. Lancet Neurol. 2013 Apr;12(4):346-56. doi: 10.1016/S1474-4422(13)70025-5. Epub 2013 Feb 26. PMID 23485610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period was form September 29, 2009 to January 19, 2011.
Pre-assignment Details: Prior to randomization, subjects needed to complete a 3-week dose adjustment of IR CD-LD followed by 6-week dose conversion to IPX066.
Groups:
- IR CD-LD (Active Comparator): Following IR CD-LD dose adjustment and conversion to IPX066, subjects were assigned to Investigational product IR CD-LD (active comparator).
Period: IR CD-LD Dose Adjustment
Arm/Group | IPX066 | IR CD-LD (Active Comparator)
Started | 0 | 471
Completed | 0 | 450
Not Completed | 0 | 21
Not completed — Adverse Event | 0 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Noncompliance with study drug | 0 | 1
Not completed — Withdrawal by Subject | 0 | 7
Not completed — Various | 0 | 9
Period: IPX066 Dose Conversion
Arm/Group | IPX066 | IR CD-LD (Active Comparator)
Started | 450 (All subjects who completed IR Dose adjustment entered into IPX066 dose conversion.) | 0 (IR is not applicable in IPX066 dose conversion.)
Completed | 393 | 0
Not Completed | 57 | 0
Not completed — Adverse Event | 23 | 0
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 13 | 0
Not completed — Withdrawal by Subject | 12 | 0
Not completed — Various | 3 | 0
Not completed — Protocol Violation | 4 | 0
Period: Maintenance - Double Blind Treatment
Arm/Group | IPX066 | IR CD-LD (Active Comparator)
Started | 201 (All subjects who completed IPX066 Dose Conversion were randomized to either IPX066 or IR.) | 192 (All subjects who completed IPX066 Dose Conversion were randomized to either IPX066 or IR.)
Completed | 186 | 182
Not Completed | 15 | 10
Not completed — Adverse Event | 3 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Noncompliance with study drug | 0 | 1
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Various | 4 | 0

BASELINE CHARACTERISTICS:
Population: All treated
Groups:
- IPX066: Investigational product IPX066
- Carbidopa-Levodopa: Immediate-release carbidopa and levodopa
- Total: Total of all reporting groups
Arm/Group | IPX066 | Carbidopa-Levodopa | Total
Number analyzed (Participants) | 201 | 192 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.0) | 63.4 (8.8) | 63.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 67 | 139
  Male | 129 | 125 | 254
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 192 | 182 | 374
  Unknown or Not Reported | 6 | 2 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  White | 196 | 186 | 382
  Black or African American | 2 | 1 | 3
  Asian | 1 | 1 | 2
  American Indian or Alaskan Native | 0 | 2 | 2
  Other | 1 | 2 | 3
  Unknown | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 8 | 18
  Romania | 3 | 4 | 7
  United States | 98 | 93 | 191
  Ukraine | 37 | 38 | 75
  Poland | 34 | 33 | 67
  France | 2 | 1 | 3
  Germany | 12 | 11 | 23
  Spain | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of "Off" Time During Waking Hours at End of Study
Description: Percentage of "off" time during waking hours at end of study is measured by using the Parkinson's disease diary. "Off" time describes a period when the participant experiences increased Parkinsonian symptoms (e.g. immobility or inability to move with ease)."
Time Frame: 22 weeks
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | IPX066 | IR CD-LD (Active Comparator)
Number analyzed (Participants) | 201 | 192
percentage | 23.82 (14.91) | 29.79 (15.81)
Statistical Analysis 1: Comparison: IR CD-LD (Active Comparator); Test type: Superiority or Other; p < .0001, ANCOVA

2. Secondary Outcome: "Off" Time
Description: "Off" time hours is measured by using the Parkinson's disease diary. "Off" time describes a period when the participant experiences increased Parkinsonian symptoms (e.g. immobility or inability to move with ease)."
Time Frame: 22 weeks
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IPX066 | IR CD-LD (Active Comparator)
Number analyzed (Participants) | 201 | 192
hours | 3.87 (2.46) | 4.88 (2.71)
Statistical Analysis 1: Comparison: IR CD-LD (Active Comparator); Test type: Superiority or Other; p < .0001, ANCOVA

3. Secondary Outcome: "On" Time Without Troublesome Dyskinesia
Description: "On" time without troublesome dyskinesiais measured by using the Parkinson's disease diary. "On" time without troublesome dyskinesia describes a period when the participant experiences decreased Parkinsonian symptoms (e.g. immobility or inability to move with ease) without dyskinesia (i.e. difficulty in performing voluntary movements) that affect daily living."
Time Frame: 22 weeks
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IPX066 | IR CD-LD (Active Comparator)
Number analyzed (Participants) | 201 | 192
hours | 11.84 (2.96) | 10.91 (2.82)

ADVERSE EVENTS:
Time Frame: 22 weeks
Arm/Group | IPX066 | Carbidopa-Levodopa
Serious Adverse Events (participants affected / at risk) | 11/201 | 5/192
Other Adverse Events (participants affected / at risk) | 57/201 | 50/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPX066 (N=201) | Carbidopa-Levodopa (N=192)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Non-cardiac Chest Pain (General disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Subdural Hematoma (Injury, poisoning and procedural complications) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine Carcinoma of the Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Acute Psychosis (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Toe Amputation (Surgical and medical procedures) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IPX066 (N=201) | Carbidopa-Levodopa (N=192)
Insomnia (Psychiatric disorders) | 7 | 2
nausea (Gastrointestinal disorders) | 6 | 3
Fall (Injury, poisoning and procedural complications) | 6 | 4
Dizziness (Nervous system disorders) | 5 | 2
Dyskinesia (Nervous system disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Oedema Peripheral (General disorders) | 4 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 4
Urinary Tract Infection (Infections and infestations) | 4 | 4
Sleep Disorder (Psychiatric disorders) | 4 | 4
Weight Decreased (Investigations) | 4 | 0
Bronchitis (Infections and infestations) | 3 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 2 | 3
On and Off Phenomenon (Nervous system disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 2 | 3
Orthostatic Hypotension (Vascular disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 4
Nasopharyngitis (Infections and infestations) | 1 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 3
Depression (Psychiatric disorders) | 1 | 5
Gait Disturbance (General disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 2
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the Study conducted at the Site shall not be made before the first multi-site publication by Sponsor.